CLINICAL TRIAL: NCT02947178
Title: Liposomal Bupivacaine Versus Bupivacaine With Fascia Iliaca Blockade for Perioperative Pain Management During Hip Arthroscopy: A Double-Blinded Prospective Randomized Control Trial
Brief Title: Hip Arthroscopy Pain Control Randomized Control Trial (RCT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 500025
Record Dates: First submitted 2016-10-12; First posted 2016-10-27 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Hip Pain Chronic; Anesthesia; Bupivacaine
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivicaine (Active Comparator): Bupivicaine fascial iliaca regional soft tissue infiltration blockade
  Interventions: Procedure: Fascial iliac regional soft tissue infiltration blockade; Behavioral: Pain Score Survey; Behavioral: Pill Count; Drug: Bupivacaine
- Bupivacaine plus liposomal bupivacaine (Active Comparator): Bupivacaine plus liposomal bupivacaine fascial iliaca regional soft tissue infiltration blockade
  Interventions: Procedure: Fascial iliac regional soft tissue infiltration blockade; Behavioral: Pain Score Survey; Behavioral: Pill Count; Drug: Bupivacaine; Drug: Liposomal Bupivacaine

INTERVENTIONS:
Procedure: Fascial iliac regional soft tissue infiltration blockade — Fascial iliac regional soft tissue infiltration blockade: Pain relief procedure (offered to all patients undergoing hip arthroscopy)
Behavioral: Pain Score Survey — Utilizing: Defense and Veterans Pain Rating Scale (DVPRS)
Behavioral: Pill Count — Patient reported as needed (prn) pain medication usage
Drug: Bupivacaine
Drug: Liposomal Bupivacaine
  Arms: Bupivacaine plus liposomal bupivacaine

SUMMARY:
Femoroacetabular impingement is a pathologic process within the hip joint that results from a mechanical discord between the femoral head and neck and the acetabulum that results in chronic hip pain, hip labral tears and early progression of osteoarthritis of the hip.1, 2 Historically an open surgical hip dislocation was performed to treat patients with this condition, however with recent advances in arthroscopy, patients more commonly now undergo arthroscopic hip surgery. From a pain management standpoint, previous attempts to provide peri-operative analgesia included intraarticular or portal analgesic injections. More recently, regional anesthesia techniques are being employed to provide more reliable and longer lasting post-operative pain control.3, 4 Currently, there are several local anesthetics available for regional anesthesia. However, they only provide an average of 12-18 hours of post-operative pain control following a single injection.5 Bupivacaine is a local anesthetic that has been used for many years by multiple routes to control post-operative pain. A new formulation of the medication prolongs the release of the active ingredient after a single injection and has been shown to result in up to 72 hours of post-operative analgesia.6, 7 To the investigator's knowledge, there has not been any studies in the literature comparing a historical control local anesthetic to this new formulation of liposomal bupivacaine via a fascial iliaca regional soft tissue infiltration blockade to provide post operative pain control following hip arthroscopy.

DETAILED DESCRIPTION:
This study is a double-blinded prospective randomized control trial. Patients will be randomized in a 1:1 ratio to either the liposomal bupivacaine group versus bupivacaine alone. Randomization assignment will be determined using a computer program based on random number generation, with an equal number of treatments in blocks of 2, 4, and 6 patients. The order of the blocks will be randomized as well. Treatment assignments will be concealed in sequentially numbered opaque sealed envelopes (SNOSE). The anesthesia provider administering the medication will not be an investigator of this study and will be allowed to know what medication that is administered to ensure safety with regards to any potential medication interactions the study medication may have with any other medication or anesthesia provided during the operation. This study will be double blinded by having the associate investigator (anesthesia resident/fellow) that will be conducting the post-operative pain score, Defense and Veterans Pain Rating Scale (DVPRS) evaluations, un-aware of which medication each patient received during the fascial iliac regional soft tissue infiltration blockade. The anesthesia resident/fellow will remain blinded to which medication the patient received by not having access to the patients electronic medical record, did not participate in the procedure, and will not have access to the database created by the orthopaedics residents where this information will be entered. The treating surgeons will also be blinded to which medication was administered by not being present during the randomization process and will only be made aware of which medication the patient received after the final two-week postoperative pain assessment and oral pain medication pill count, after which patient study participation will be concluded. The success of blinding will be evaluated by asking the patient, anesthesia resident/fellow and treating surgeon to guess their treatment assignment the day of surgery, during the pain score collection process and at the final two-week routine follow up appointment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is scheduled to undergo hip arthroscopy
2. Patient is between 18-50 years of age
3. DEERS eligibility

Exclusion Criteria:

1. Patients who are on a medication pre-operatively that would prohibit them from receiving one of the study medications
2. Patient is unable to speak/read the English language (Currently, the DVPRS has only been scientifically validated in the English language and translating to languages other than English would compromise the validity of the pain scale)
3. Patient has a history of previous hip arthroscopy surgery
4. The patient is pregnant - ruled out with routine urine pregnancy test the morning of surgery in the anesthesia pre-operative unit.
5. The patient carries a pre-existing diagnosis of a pain disorder. (Example: Fibromyalgia)
6. The patient has a previous history of narcotic pain medication abuse.
7. The patient has an allergy to one of the study medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Pain | Immediate Post-operative
  To compare post-operative pain scores between the two treatments groups. To advance this objective, DVPRS (Defense and Veterans Pain Rating Scale) scores will be collected and analyzed at discharge and on post-operative days one, two, and three. The investigator's hypothesize that the addition of liposomal bupivacaine will result in a 2-point improvement in DVPRS scores during the post-operative period.

SECONDARY OUTCOMES:
Opioid Use | Immediate Post-operative
  To compare overall post-operative opioid use between the two treatment groups. Opioid usage will be quantified using a patient-reported medication diary and a pill count. The investigator's hypothesize that the addition of liposomal bupivacaine will result in a decrease in total opioid use during the post-operative time period.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kent, MD, Study Director — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be combined together for data analysis.